CLINICAL TRIAL: NCT01696617
Title: Aripiprazole (Abilify®) as an Adjunctive Treatment for Inadequate Response in Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yong Min Ahn, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 031-KOC-1108i
Record Dates: First submitted 2012-07-31; First posted 2012-10-01 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Aripiprazole; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aripiprazole 8-week group (Experimental): Adjunctive aripiprazole 8-week treatment
  Interventions: Drug: Aripiprazole 6-week group
- Aripiprazole 6-week group (Active Comparator): Adjunctive aripiprazole 6-week treatment
  Interventions: Drug: Aripiprazole 8-week group

INTERVENTIONS:
Drug: Aripiprazole 6-week group
  Other Names: Abilify®
  Arms: Aripiprazole 8-week group
Drug: Aripiprazole 8-week group
  Other Names: Abilify®
  Arms: Aripiprazole 6-week group

SUMMARY:
The investigators hypothesized that combined pharmacotherapy using adjunctive aripiprazole of standard antidepressants would be associated with improved depression response in Major depressive disorder, especially in Quality of life.

The investigators compare the mean changes in the quality of life between before add-on and 8 weeks treatment of aripiprazole and between before add-on and 6 weeks treatment of aripiprazole.

DETAILED DESCRIPTION:
Previous study about quality of life measurement in patients with depression have been reported that quality of life have to be measured irrespective with the severity of depression because quality of life has some other aspect to depression.The investigators have designed a 6-week single blinded study with flexible dose aripiprazole augmentation, ranging from 2.5mg to maximum 20 mg (15mg for patients on fluoxetine or paroxetine), in patients who responded inadequately (a score of >18 on the MADRS) to first-line antidepressant pharmacotherapy. The investigators compare the mean changes from in the quality of life at 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age : 18-65
* Patients with major depressive disorder according to DSM-IV criteria that have lasted >8 weeks
* MADRS total score of 18 or higher
* Patients who responded inadequately (a score of >18 on the MADRS) to first-line antidepressant treatment of 4 week duration
* Current use of standard antidepressant treatment in monotherapy or combination of 2 antidepressants : escitalopram (10 - 20mg/d), fluoxetine(20 - 40mg/d), paroxetine CR(25 - 50mg/d), sertraline(100 - 150mg/d), mirtazapine (15 - 45mg/d), duloxetine (30 - 60mg/d) or venlafaxine ER(150-225mg/d)

Exclusion Criteria:

* Past history of hypersensitivity to aripiprazole
* Primary diagnosis of MDD with psychotic feature, bipolar disorder, schizophrenia, schizoaffective disorder, other psychotic disorder or anxiety disorder, a history of alcohol/ drug abuse within the past 12 months, or a diagnosis of dementia
* Clinically significant current Axis II (DSM-IV-TR) diagnosis
* A significant risk of suicide corroborated by a score of ≥5 on item 10(suicidal thoughts) on the MADRS scale or by clinical judgment of the investigator
* Pregnancy or in breast-feeding
* Presence of a serious medical illness including cardiac, hepatic, renal, respiratory, endocrinologic, neurologic, or hematologic disease or physical disorder judged to significantly affect central nervous system function
* Patients taking antipsychotics, mood stabilizer or any psychotropic medications besides antidepressants, except benzodiazepines or beta blockers or hypnotics
* Patients with past treatment failures of aripiprazole

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-02-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Quality of Life Scale (QOLS) | Change from Baseline at 8 weeks
  change of Quality of Life Scale (QOLS)

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale | Change from Baseline at 8 weeks
  change of Montgomery-Åsberg Depression Rating Scale

OTHER OUTCOMES:
Hamilton Rating Scale for Depression | Change from Baseline at 8 weeks
  change of Hamilton Rating Scale for Depression
Clinical Global Impression-severity, Clinical Global Impression-Improvement | Change from Baseline at 8 weeks
  change of Clinical Global Impression-severity, Clinical Global Impression-Improvement
Beck Depression Inventory | Change from Baseline at 8 weeks
  change of Beck Depression Inventory
Inventory of Depressive Symptomatology Self-Report Scale | Change from Baseline at 8 weeks
  change of Inventory of Depressive Symptomatology Self-Report Scale
Drug - Induced Extrapyramidal Symptoms Scale | Change from Baseline at 8 weeks
  change of Drug - Induced Extrapyramidal Symptoms Scale
The Liverpool University Neuroleptic Side Effect Rating Scale | Change from Baseline at 8 weeks
  change of The Liverpool University Neuroleptic Side Effect Rating Scale
Short From-36 Health survey | Change from Baseline at 8 weeks
  change of Short From-36 Health survey

CONTACTS AND LOCATIONS:
Overall Officials: Yong Min Ahn, MD. Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea